CLINICAL TRIAL: NCT01226628
Title: Phase 1/2a, Multicenter, Randomized, Dose Escalation, Fellow-Eye Controlled, Study Evaluating the Safety and Clinical Response of a Single, Subretinal Administration of Human Umbilical Tissue-Derived Cells (CNTO 2476) in Subjects With Visual Acuity Impairment Associated With Geographic Atrophy Secondary to Age-related Macular Degeneration
Brief Title: A Safety Study of CNTO 2476 in Patients With Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017548; CNTO2476MDG1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Age-related Macular Degeneration
Keywords: Macular degeneration; Age-related macular degeneration; Cell therapy; CNTO 2476; Human umbilical tissue-derived cells; hUTC; Geographic Atrophy; Subretinal; Visual Acuity
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort A (Experimental): Phase 1: 3 patients will receive 60,000 human umbilical tissue-derived cells (hUTC)
  Interventions: Biological: CNTO 2476; Procedure: iTrack Model 275 micro catheter
- Cohort B (Experimental): Phase 1: 3 patients will receive 120,000 hUTC
  Interventions: Biological: CNTO 2476; Procedure: iTrack Model 275 micro catheter
- Cohort C (Experimental): Phase 1: 3 patients will receive 300,000 hUTC
  Interventions: Biological: CNTO 2476; Procedure: iTrack Model 275 micro catheter
- Cohort D (Experimental): Phase 1: 3 patients will receive 560,000 hUTC
  Interventions: Biological: CNTO 2476; Procedure: iTrack Model 275 micro catheter
- Cohort E (Experimental): Phase 1: 6 patients will receive 300,000 hUTC
  Interventions: Biological: CNTO 2476; Procedure: iTrack Model 275 micro catheter
- Cohort F (Experimental): Phase 1: 6 patients will receive either 60,000 or 300,000 hUTC
  Interventions: Biological: CNTO 2476; Procedure: iTrack Model 275 micro catheter
- Cohort G (Experimental): Phase 1: 6 patients will receive either 60,000 or 300,000 hUTC
  Interventions: Biological: CNTO 2476; Procedure: iTrack Model 275 micro catheter
- Phase 2a (Experimental): Up to 38 patients will receive one of two optimal doses as selected from the Phase 1 portion of the study
  Interventions: Biological: CNTO 2476; Procedure: iTrack Model 275 micro catheter

INTERVENTIONS:
Biological: CNTO 2476
  Other Names: Palucorcel
Procedure: iTrack Model 275 micro catheter — CNTO 2476 will be administered subretinally using the iTRACK microcatheter in participants with visual acuity impairment. During surgery, the portion of microcatheter distal to the flexible blue hub is inserted into the subretinal space via a peripheral scleral cutdown and choroidal fistula.

SUMMARY:
The main purpose of this study to evaluate the safety and tolerability of CNTO 2476 administered subretinally (beneath the retina) using the iTrack Model 275 micro catheter in patients with visual acuity (acuteness or clearness of vision) impairment associated with the geographic atrophy (GA: partial or complete wasting away of retinal layer below the retina) manifestation of age-related macular degeneration (AMD: medical condition which usually affects older adults and results in a loss of vision in the center of the visual field [the macula] because of damage to the retina).

DETAILED DESCRIPTION:
The study is a Phase 1/2a, multicenter, randomized (the study medication is assigned by chance), single dose, dose escalation, fellow-eye controlled study evaluating the safety and clinical response of a single, subretinal administration of CNTO 2476 in patients with visual acuity impairment associated with GA secondary to AMD. The study will consist of screening (up to 21 days prior to treatment) period, treatment (Day 1) period and follow up period. The study will be conducted in 2 portions: the Phase 1 portion will include dose escalation and the Phase 2 portion will enroll additional patients randomized to one of the 2 optimal doses selected from the Phase 1 portion (with an acceptable safety profile seen in Phase 1). For Phase 1, the treatment eye will be the eye with worse visual acuity or the one chosen by the investigator, however, the treatment eye cannot have a visual acuity no better than 20/200. For Phase 2a, the treatment eye will be the eye with worse visual acuity, and cannot have a visual acuity better than 20/80. Approximately 30 patients will participate in the Phase 1 dose escalation portion, and 38 patients will be enrolled in the Phase 2a portion (19 patients receiving optimal dose level X from Phase 1 and 19 receiving optimal dose level Y from Phase 1). In the Phase 1 portion, treatment will be assigned 5 sequential cohorts, with 3 patients per cohort in each of the first 4 cohorts and 6 patients in the fifth cohort. Cohort A patients will be treated first, followed by Cohort B patients. All patients in a given cohort must have completed at least 4 weeks of post-treatment follow-up before patients in the next cohort may be treated. Follow-up will include postoperative follow-up period of 12 months (Day 2, Day 7, Day 15, Week 3, Week 4, Months 2, 3, 6, and 12) and long-term safety follow-up period (patients will be evaluated every 6 months for safety assessments). Safety assessments will include vital signs, AEs, and concomitant medications and routine 12-lead electrocardiograms (ECG). The anticipated study duration will be approximately 5 years (1 year in the 12-month postoperative follow-up period; up to 4 years in the long-term safety follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* Women must be incapable of childbearing
* Patient must be a suitable candidate for ophthalmologic surgery, is willing and able to comply with the surgical procedure, scheduled visits, treatment plan, laboratory tests and other study procedures
* Confirmed diagnosis of bilateral geographic atrophy (GA) of the macula bilaterally caused by age-related macular degeneration

Exclusion Criteria:

* Evidence of exudative ("wet") age -related macular degeneration in either eye
* Evidence of other significant ophthalmologic disease (eg, glaucoma)
* Ocular hypertension
* Previous cell therapy other than blood components
* Previous treatment for age-related macular degeneration (AMD) other than antioxidant or zinc supplements or other oral vitamin supplements

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-10-21 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Number of eyes with serious ocular adverse events occurring over the first 12 months of the study | 12 months
  This number will be summarized descriptively for treated and fellow eyes within each dose level included in Phase 1 and Phase 2a portions of the study

SECONDARY OUTCOMES:
Change from baseline in antibody peak values | Baseline (Screening), up to 60 months
Yearly rate of increase from baseline in area of Geographic Atrophy (GA) | Baseline (Screening), up to 60 months
Changes from baseline in visual function | Baseline (Screening), up to 60 months
  Changes from baseline in visual function is measured as changes in best corrected visual acuity [BCVA], low luminance BCVA, low luminance deficit, reading speed, contrast threshold, visual field and retinal thickness measured by spectral-domain optical coherence tomography (SD-OCT) at registered sections of the macula that include the geographic atrophy and adjacent retina
Change from baseline in Visual Functioning Questionnaire (VFQ)-25 | Baseline (Screening), up to 60 months
  The VFQ-25 is a reliable and validated 25-item version of the larger 51-item National Eye Institute Visual Function Questionnaire. The questionnaire must be administered by the study staff and must not be self-administered. Analysis of VFQ-25 questionnaire data will be based on the thirteen sub-scales and a composite score.
Incidence of adverse events | up to 60 months
  Incidence of adverse events will be assessed in both Phases (Phase 1 and Phase 2a)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Arcadia, California
  - Philadelphia, Pennsylvania